CLINICAL TRIAL: NCT01492803
Title: A Randomized Placebo-Controlled Trial of Probiotics to Lower Microbial Translocation and Immune Activation in HIV-Infected Adolescents
Brief Title: Trial of Probiotics to Lower Microbial Translocation and Immune Activation in HIV-Infected Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ATN 097
Record Dates: First submitted 2011-11-04; First posted 2011-12-15 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: HIV infection; Probiotics
MeSH Terms: conditions — HIV Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm.
  Interventions: Dietary Supplement: Placebo
- Probiotics (Experimental): The probiotics use in the study contains two strains of Lactobacillus plantarum. Each dose of the active study agent contains contains 1 g maltodextrin plus the probiotic bacteria Lp299v (5 x 109 cfu) and Lp299 (5 x 109 cfu).
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotic is a live microorganism that when administered in adequate amounts confer a health benefit on the host. It is classified by the FDA as "generally recognized as safe" (GRAS)
  Other Names: No other names.
  Arms: Probiotics
Dietary Supplement: Placebo — The placebo sticks will contain approximately 1 g maltodextrin
  Arms: Placebo

SUMMARY:
This is a randomized placebo-controlled trial to examine if once daily probiotic therapy will lower serum LPS levels and immune activation among HIV-infected youth.

DETAILED DESCRIPTION:
This is a double masked randomized placebo-controlled trial to examine if once daily probiotic therapy will lower serum lipopolysaccharide (LPS) levels and immune activation among HIV-infected youth. The study will enroll two cohorts: (1) a cohort of subjects who are not receiving antiretroviral therapy (ART) and have absolute CD4 T-cell count greater than 350 cells/ul and quantitative HIV-1 plasma RNA (viral load) less than 50,000 copies/ml; and (2) a cohort of subjects who are receiving ART and have absolute CD4 T-cell count greater than 350 cells/ul and and quantitative HIV-1 plasma RNA (viral load) less than 400 copies/ml.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment, an individual must meet the criteria listed below.

* Age 13 years and 0 days to 24 years and 364 days at the time of consent
* Confirmed or suspected to have acquired HIV infection at age 10 years or older
* HIV-1 infection as documented by any FDA-approved ELISA test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, HIV-1 DNA, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA at any time prior to pre-entry
* Absolute CD4 T-cell count greater than 350 cells/ul at pre-entry
* Cohort 1 - Not receiving ART and no exposure to ART in the 24 weeks prior to pre-entry: Quantitative HIV-1 plasma RNA (viral load) less than 50,000 copies/ml on two consecutive determinations at least 8 weeks apart in the 24 weeks prior to and including pre-entry
* Cohort 2 - Currently receiving ART and received ART for at least the 24 weeks prior to pre-entry: Quantitative HIV-1 plasma RNA (viral load) less than 400 copies/ml on two consecutive determinations at least 8 weeks apart in the 24 weeks prior to and including pre-entry
* Willingness to refrain from regular use of foods/supplements containing probiotics other than that supplied by the study during the course of study participation

Exclusion Criteria:

To be considered eligible for enrollment, an individual must not meet any of the criteria listed below.

* Known hypersensitivity to probiotics
* Active AIDS-defining condition or acute serious illness
* Cohort 1 - Not receiving ART and no exposure to ART in the 24 weeks prior to pre-entry: Any quantitative HIV-1 plasma RNA (viral load) equal to or greater than 50,000 copies/ml during the 24 weeks prior or at pre-entry.
* Cohort 2 - Currently receiving ART and received ART for at least the 24 weeks prior to pre-entry: Any quantitative HIV-1 plasma RNA (viral load) equal to or greater than 400 copies/ml during the 24 weeks prior or at pre-entry
* Known history of inflammatory bowel disease or similar disorder of the GI tract
* Current treatment with immune-modulating or immune-suppressive therapy
* Active malignancy at pre-entry
* Pregnancy
* Grade 3 or higher clinical or laboratory toxicities at the time of randomization
* Regular use of foods or supplements containing probiotics within the 2 weeks prior to randomization (see Appendix V)
* Concurrent participation in the ATN 061, 071, 081, and/or 101 protocols

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Plasma LPS levels | 32 Weeks
  To determine if once daily probiotic therapy decreases microbial translocation in HIV-infected youth as measured by changes in plasma LPS.

SECONDARY OUTCOMES:
Stool colonization with Lactobacillus plantarum | 32 Weeks
  To quantify the extent that Lactobacillus plantarum populates fecal samples obtained over time in HIV-infected youth receiving probiotics.
Plasma pro-inflammatory cytokines and macrophage activation | 32 Weeks
  To determine if probiotic colonization of the gastrointestinal (GI) tract with Lactobacillus plantarum decreases levels of plasma pro-inflammatory cytokines and macrophage activation by measuring tumor necrosis factor alpha (TNFα), interferon alpha (IFNα), interleukin-1 beta (IL-1β), interleukin-6 (IL-6), interleukin-12p70 (IL-12p70), interleukin-10 (IL-10), and soluble CD14 (sCD14) as well as other markers of microbial translocation.
Lymphocyte activation markers | 32 Weeks
  To determine if probiotic colonization of the GI tract with Lactobacillus plantarum results in decreased levels of T-cell activation markers as measured by shedding of soluble CD27 (sCD27), proportion of CD4 Th17 subsets, and expression of CD38 and HLA DR on CD8 T cells within ART treated and untreated HIV-infected youth.
Quantitative HIV-1 plasma RNA (viral load) and CD4 T-cell count | 32 Weeks
  To examine if probiotics have any impact on quantitative HIV-1 plasma RNA (viral load) and CD4 T-cell count among the study cohort.
Stool microbial composition and genetic diversity | 32 Weeks
  To molecularly characterize changes in overall bacteria diversity within the stool specimens of youth treated with probiotics.
Safety labs and adverse events as a measure of acceptability and tolerability of probiotics | 32 Weeks
  To examine the acceptability and tolerability of probiotics when administered to HIV-infected youth.
Food frequency and probiotics and lifestyle questionnaires | 32 Weeks
  To explore the effect of diet, smoking, and dietary supplements on plasma pro-inflammatory cytokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: John Sleasman, MD, Study Chair — University of South Florida

REFERENCES:
- See also: ATN website — http://atnonline.org